CLINICAL TRIAL: NCT04905238
Title: Pathophysiology Consequences of Obstructive Sleep Apnea in Biomarkers of Alzheimer's Disease. A Clinical Trial
Brief Title: Obstructive Sleep Apnea and Biomarkers of Alzheimer's Disease
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Alberto Alonso Fernandez (Other Government)
Collaborators: Instituto de Salud Carlos III (Other Government)
Responsible Party: Sponsor-Investigator, Alberto Alonso Fernandez, Principal investigator, Fundació d'investigació Sanitària de les Illes Balears
Organization: Fundació d'investigació Sanitària de les Illes Balears (Other Government)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AOS-AD
Record Dates: First submitted 2021-05-24; First posted 2021-05-27 (Actual); Last update posted 2025-05-01 (Actual); Status verified 2025-04

CONDITIONS: Sleep Apnea, Obstructive
Keywords: sleep apnea obstructive
MeSH Terms: conditions — Sleep Apnea, Obstructive | interventions — Continuous Positive Airway Pressure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Continuous positive airway pressure (Active Comparator): Diet and general life style recommendations plus continuous positive airway pressure (CPAP).
  Interventions: Device: Continuous positive airway pressure
- Conservative treatment (No Intervention): Diet and general life style recommendations.

INTERVENTIONS:
Device: Continuous positive airway pressure — Continuous positive airway pressure
  Arms: Continuous positive airway pressure

SUMMARY:
Clinical trial on the effect of continuous positive pressure (CPAP). Objectives: 1) To compare biomarkers of Alzheimer's disease in plasma samples from patients with Obstructive sleep apnea (OSA) and without OSA. 2) To determine if CPAP reduces biomarkers of Alzheimer's disease in plasma samples.

DETAILED DESCRIPTION:
Randomized, parallel group, non-blinded, controlled clinical trial compared with conventional treatment.

A. Protocol and intervention Patients with an Apnea-Hypopnea index (AHI)>30 h-1 will be assigned, using a 1:1 randomization table, to lifestyle recommendations treatment or to lifestyle recommendations plus nasal CPAP, for a period of 4 months. CPAP pressure will be titled with automatic using an AutoSet II device, ResMed.

B. Sample size For the estimation of the sample size, previous data were used (PLoS ONE 2019;14(9): e0221255). In this case, in order to compare the effect of CPAP it would be necessary to randomize a total of 100 patients with OSA and 30 control subjects.

C. Ethical considerations

* Indication of CPAP treatment for the prevention of Alzheimer's disease is not yet accepted.
* Those patients with an urgent study indication for the diagnosis and treatment of respiratory sleep disorders (professional drivers, respiratory failure or risk professions) will be excluded from the project. In the other cases, the delay in healthcare for the performance of Polysomnography and CPAP titration exceeds the duration of the study, therefore that patients assigned to the control arm (conventional treatment) will not be exposed to a higher risk than the general population.

D. Methods.

. Polysomnography. It will be used as a screening test previous the randomization of the included patients. The exploration and its interpretation will be carried out following the recommendations of the American Academy of Sleep Medicine. Based on the results of this test, only those patients with an AHI will continue in the study when AHI >30 h-1. In these patients the determinations listed below will be carried out immediately before randomization (visit 1), at 4 weeks (visit 2), 16 weeks (visit 4) of allocation to the corresponding treatment group

* Clinical data: The medication used and other associated diseases already diagnosed will be recorded.
* Vital signs: recording of blood pressure, by means of a conventional triple taking, and heart rate.
* Anthropometric characteristics: age and weight in basal conditions, the perimeter of the neck and waist / hip index will be measured. The lean mass index will be determined using a Bodystat 1500 impedance system (Bodystat Ltd, United Kingdom).
* Questionnaires: Epworth Sleepiness Scale, generic health-related quality of life (SF-12 and EuroQoL) and daily physical activity (International Physical Activity Questionnaire or iPAQ).
* Laboratory findings: blood count, coagulation, creatinine, serum sodium and potassium; glycated hemoglobin (HbA1c) and blood glucose and insulin levels in fasting, from these values will determine the resistance and sensitivity to insulin using the homeostatic model assessment (HOMA) and Quantitative insulin sensitivity check index (QUICKI) indices; total cholesterol, HDL-cholesterol, LDL-cholesterol and triglycerides; and troponin I, homocysteine, N-terminal pro-brain natriuretic peptide (NT-pro BNP) and highly sensitive C-reactive protein.
* Blood venous samples. 20 mL of venous blood will be collected, storing the plasma obtained at -80 ºC for subsequent determination of β amyloid biomarkers (Aβ40, Aβ42, tau y tau 181 (P-tau 181).
* Night pulse oximetry. To assess the existence of residual nocturnal hypoxemia.
* In the patients assigned to the CPAP treatment arm, a count of the hours of use of the CPAP will be carried out at each visit by directly reading the automatic counter of each equipment.

Statistic analysis The data will be expressed as mean ± standard deviation, median (interquartile range) or percentage, depending on their type and distribution. For comparison between groups Student's t-test, the U-Mann-Whitney or the chi-square test will be used, as appropriate. The relations between variables will be analyzed using Pearson's correlation and multiple linear regression analysis. The effect of treatment will be evaluated using general linear models and repeated measures analysis of variance, with multiple comparisons post-hoc using the Bonferroni test. A multiple logistic regression model will be applied to determine the related variables with a response to treatment. Values of p <0.05 will be considered statistically significant. The statistical study will be performed with the SPSS program version 22.0.

ELIGIBILITY:
Inclusion Criteria:

* Cases: patients with AHI > 30/h
* Controls: subjects with AHI < 5/h and Epworth <10

Exclusion Criteria:

* Epworth>18
* BMI<40Kg/M2
* Arterial Hypertension
* Diabetes Mellitus
* Cerebrovascular disease
* Ischemic heart disease
* Cardiac arrhythmia
* Chronic cardiovascular diseases
* Daytime Oxygen saturation>95%
* Risk professions (professional drivers)
* Concomitant treatment with antihypertensives, statins, antidiabetics, beta- blockers or systemic corticosteroids.
* Pretreatment with CPAP.
* Participation in another clinical trial thirty days prior to randomization
* Abnormal values of a cognitive test.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2020-07-31 (Actual); Primary Completion 2025-04-10 (Actual); Study Completion 2025-05-06 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in β-amyloid 40 (Aβ-40 and/or Aβ42) concentration | 4 months
  To compare the change in Aβ-40 and/or Aβ42 levels between the patients allocated to CPAP group and the control group
β-amyloid 40 (Aβ-40 and and/or Aβ42) concentration in OSA and in non-OSA patients | Baseline
  To compare Aβ-40 and/or Aβ42 levels between OSA and non-OSA patients

SECONDARY OUTCOMES:
Phospho-Tau (P-Tau) concentration in OSA and in non-OSA patients | Baseline
  To compare plasma concentrations of P-Tau in subjects with/without OSA.
Apolipoprotein E (APOE) concentration in OSA and in non-OSA patients | Baseline
  To compare plasma concentrations of Apolipoprotein E (APOE) in subjects with/without OSA.
Neurofilament light chain (NfL) concentration in OSA and in non-OSA patients | Baseline
  To compare plasma concentrations of NfL in subjects with/without OSA.
Microbiota population diversity from stool and nasopharyngeal samples in OSA and in non-OSA patients | Baseline
  To compare microbiota population diversity from stool and nasopharyngeal samples in OSA and in non-OSA patients
Microbiota population abundance from stool and nasopharyngeal samples in OSA and in non-OSA patients | Baseline
  To compare microbiota abundance from stool samples and nasopharyngeal samples in OSA and in non-OSA patients
Microbiota population color maps from stool and nasopharyngeal samples in OSA and in non-OSA patients | Baseline
  To compare microbiota population color maps from stool and nasopharyngeal samples in OSA and in non-OSA patients
Associations of microbiota population diversity from stool and nasopharyngeal samples in OSA with biomarkers of Alzheimer's Disease | Baseline
  To relate microbiota population diversity from stool and nasopharyngeal samples to biomarkers of Alzheimer's Disease
Associations of microbiota population abundance from stool and nasopharyngeal samples in OSA with biomarkers of Alzheimer's Disease | Baseline
  To relate microbiota population abundance from stool and nasopharyngeal samples to biomarkers of Alzheimer's Disease
Associations of microbiota population color maps from stool and nasopharyngeal samples in OSA with biomarkers of Alzheimer's Disease | Baseline
  To relate microbiota population color maps from stool and nasopharyngeal samples to biomarkers of Alzheimer's Disease
To evaluate the relationship of biomarkers of Alzheimer's disease and oropharyngeal and gut microbiota with the main classical markers of OSA and nocturnal hypoxic burden. | Baseline
  To evaluate the relationship of biomarkers of Alzheimer's disease and oropharyngeal and gut microbiota with the main classical markers of OSA (AHI, AHI in REM, Di, arousals index, slow wave sleep time, SpO2 time<90%, mean nocturnal SpO2, minimum SpO2, 3% and 4% desaturations index), as well as with nocturnal hypoxic burden related to respiratory events.
Associations between CPAP effects on oropharyngeal and gut microbiota, and biomarkers of Alzheimer's disease. | 4 months
  To assess whether CPAP treatment modifies microbiota population diversity, abundance, and color maps from stool samples and nasopharyngeal samples of patients with OSA, and whether these changes correlate with variations in biomarkers of Alzheimer's disease
Change from baseline in biomarkers of Alzheimer's disease, and oropharyngeal and gut microbiota samples of patients with OSA according to the baseline hypoxic burden level and residual hypoxia. | 4 months
  To assess whether residual hypoxia and baseline hypoxic burden results in a different response to CPAP/conservative treatment on biomarkers of Alzheimer's disease, and oropharyngeal and gut microbiota in patients with OSA.
To determine the relationship between compliance with CPAP treatment and the response on biomarkers of Alzheimer's disease and oropharyngeal and gut microbiota. | 4 months
  To assess whether CPAP compliance (>4 hours) results in a different response to biomarkers of Alzheimer's disease, and oropharyngeal and gut microbiota in patients with OSA.

CONTACTS AND LOCATIONS:
Locations (2):
- Spain (2):
  - Hospital Son Espases, Palma, Balearic Islands
  - Hospital Son Llatzer, Palma, Balearic Islands